CLINICAL TRIAL: NCT00969592
Title: Comparison of Pharmacodynamics and Pharmacokinetics of the Two Fast-acting Insulin Analogs Insulin Glulisine and Insulin Aspart in Healthy Volunteers
Brief Title: Expanded PK and PD of Insulin Glulisine Versus Insulin Aspart in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Christoph Kapitza, MD, Profil Institut für Stoffwechselforschung GmbH
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 49-0361-GluAsp
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin glulisine; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin glulisine, insulin aspart (Active Comparator): insulin glulisine administration during first glucose clamp, insulin aspart administration during second glucose clamp
  Interventions: Drug: insulin glulisine, insulin aspart
- insulin aspart, insulin glulisine (Active Comparator): insulin aspart administration during first euglycemic clamp, insulin glulisine administration during second clamp
  Interventions: Drug: insulin aspart, insulin glulisine

INTERVENTIONS:
Drug: insulin glulisine, insulin aspart — single subcutaneous dose of 0.2 units per kg body weight of insulin glulisine during first euglycemic glucose clamp, single subcutaneous dose of 0.2 units per kg body weight of insulin aspart during second euglycemic glucose clamp
  Other Names: Apidra; NovoRapid
  Arms: insulin glulisine, insulin aspart
Drug: insulin aspart, insulin glulisine — single subcutaneous dose of 0.2 units per kg body weight of insulin aspart during first euglycemic glucose clamp, single subcutaneous dose of 0.2 units per kg body weight of insulin glulisine during second euglycemic glucose clamp
  Other Names: NovoRapid; Apidra
  Arms: insulin aspart, insulin glulisine

SUMMARY:
The purpose of this study was to compare the pharmacodynamics (course of the blood glucose-lowering effect and duration of effect) and pharmacokinetics (course of the concentration of study medication in the blood) of a single subcutaneous dose of 0.2 units/kg of insulin glulisine and insulin aspart in a direct head-to-head comparison during two euglycemic glucose clamps in healthy subjects.

DETAILED DESCRIPTION:
In a previous glucose clamp study with a head-to-head comparison of insulin glulisine and insulin lispro it was shown that the onset of metabolic action was significantly shorter with insulin glulisine than with insulin lispro (while the total metabolic effect was not different). These results were in line with a faster early insulin exposure of insulin glulisine compared to insulin lispro. The primary aim of this study was to investigate whether or not these favorable characteristics of insulin glulisine were also evident in the comparison against insulin aspart. This was the first clinical study realizing a head-to-head comparison between these two insulin analogs.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females (Women: contraception, Pearl Index <1%)
* Between the ages of 18 and 65 years
* Body Mass Index of <= 27 kg/m²
* Safety lab within reference range
* Normal blood pressure and heart rate
* Sufficient venous access
* Written informed consent approved by the Ethical Review Board
* HbA1c and fasting plasma glucose in the normal range

Exclusion Criteria:

* Investigative site personnel directly affiliated with this study and their immediate families or the sponsor´s employees
* Within 30 days of the initial dose of study drug had received treatment with a drug that had not received regulatory approval
* Known allergies to insulin or related compounds
* Regular treatment with any drug, both over-the-counter or prescribed
* an abnormality in the 12-lead ECG increasing the risk for participation
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Significant active neuropsychiatric disease
* Regular use of drugs of abuse and or positive findings on urinary drug screening
* Evidence of HIV and/or positive antibodies 1 or 2 and or HIV1 antigen
* Evidence of hepatitis B and/or positive hepatitis C antibody
* Evidence of hepatitis B and/or positive hepatitis B surface antigen
* Women with a positive pregnancy test or breastfeeding women
* Blood donation more than 500 mL within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
fractional and total glucose infusion rates | 0-1 hours, 0-2 hours, and time to 10% of GIRmax

SECONDARY OUTCOMES:
fractional and total insulin areas under the curve (AUC) | 0-1 hours, 0-2 hours, 0-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Arnolds, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany